CLINICAL TRIAL: NCT01679340
Title: Phase Ⅱ Study of S-1 Combined With Oxaliplatin (SOX)Verse S-1 Combined With Cisplatin(SP) in Adjuvant Chemotherapy After D2 Surgery
Brief Title: A PhaseⅡ Study: SOX vs SP in Adjuvant Chemotherapy After D2 Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shen Lin, Director of GI oncology, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SOXSP
Record Dates: First submitted 2012-06-13; First posted 2012-09-06 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; D2 surgery; S-1; Oxaliplatin; cisplatin
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); titanium silicide; Oxaliplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S-1+oxaliplatin (Experimental): S-1: 80mg/m2, 3weeks/cycle(take for 14d, rest for 7d oxaliplatin: 65mg/m2, D1,D8, 3weeks/cycle after 6 cycles, then mono S-1 for 2-4 cycles, total 8-10 cycles.
  Interventions: Drug: S-1; Drug: oxaliplatin
- S-1+cisplatin (Active Comparator): S-1: 80mg/m2, 3weeks/cycle(take for 14d, rest for 7d) cisplatin: 75mg/m2, D1, every 3 weeks After 6 cycles, then mono S-1 for 2-4 cycles, total 8-10 cycles.
  Interventions: Drug: S-1; Drug: cisplatin

INTERVENTIONS:
Drug: S-1 — Mode of administration: orally (capsules) Dosing schedule:80mg/m2, Bid,D1-14,every 3 week,for 8-10cycles
  Other Names: TS-1; Aisiwan
Drug: oxaliplatin — Mode of administration: intravenously Doseing schedule: 65 mg/m2 D1,D8,every 3 week, for 6 cycles
  Arms: S-1+oxaliplatin
Drug: cisplatin — Mode of administration: intravenously Dosing schedule: 75mg/m2 D1,every 3 week,for 6 cycle
  Arms: S-1+cisplatin

SUMMARY:
To investigate the efficiency and safety of SOX or SP adjuvant chemotherapy to phase II and III gastric cancer patients after D2 surgery. If SOX is equal to SP in efficiency and less toxicity.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed Phase III adenocarcinoma of gastric and esophageal-gastric junction ( AJCC 7th)
* without previous treatment, including radiotherapy, chemotherapy and immunotherapy
* Hb≥90g/L,WBC 4×109/L-10×109/L,ANC≥2×109/L,Platelet≥100×109/L
* creatinine≤1 UNL
* total bilirubin≤1.5 UNL,AST(SGOT),ALT(SGPT) and ALP≤2.5 UNL
* ECOG score 0 - 2
* take chemotherapy for 8 weeks after surgery
* older than 18 years
* can be followed up, good compliance
* can take medicine orally
* having signed informed consent

Exclusion Criteria:

* combined disease lead to Life Expectancy less than 3 years
* any evidence to show metastasis,including cancer cells in peritoneal fluid
* inability to take oral medication for difficult to swallow, intestinal obstruction，active intestinal blooding or perforation
* previous treatment,including cytotoxic chemotherapy, radio chemotherapy or immunotherapy ( except corticosteroid hormone）
* operation within 4 weeks, or not recovered from last major operation
* allergy with fluorouracil
* allergy with Platinum or any composition in research drugs
* uncontrollable seizure disorder，central nervous system disease or mental disorders, and has clinical significance by judgement of researchers, or can influnce understanding of informed consent or compliance to take orally drugs
* in the past 12 months, has clinical significant heart disease(active),such as symptomatic coronary heart disease, > =Stage II congestive cardiac failure;congestive heart failure as NYHA standard, or serious arrhythmias need take medicine( as Appendix 10th),or myocardical infarction.
* pregnancy， lactation， women in child-bearing period and her spouses reject to take effictive method to conraception
* other previous malignancy within 5 years, except healed skin basal cell carcinoma and carcinoma in cervix
* peripheral neuropathy> grade 1 of CTCAEv3, except the neural abnormality patients who only lose deep tendon reflex（DTRs）.
* serious complicated infection or other complicated diseases and hard to controll.
* As one of belowing:
* ANC < 2×109/L
* Platelet<100×109/L
* total bilirubin>1.5 UNL
* ALAT、ASAT > 2.5 x ULN
* ALP> 2.5 x ULN
* Any investigational agent within the past 28 days. That is the patient had jioned another trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-04; Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
replase free survival | 3 months

SECONDARY OUTCOMES:
overall survival | 6 months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China